CLINICAL TRIAL: NCT06851130
Title: Assessing the Immediate Increase in Serum Ferritin After Oral Iron Doses: an Experimental Study in Iron-deficient Women
Acronym: INFER 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INFER Study 2
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Iron Deficiency Without Anemia
Keywords: serum ferritin; oral iron supplementation
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 80 mg (Experimental): Daily dose of 80 mg of iron for 1 month, with a 7-day break, then again for another month (2 months total).
  Interventions: Dietary Supplement: ferrous sulfate 80 mg
- 160 (Experimental): Daily dose of 160 mg of iron for 1 month, with a 7-day break, then again for another month (2 months total).
  Interventions: Dietary Supplement: ferrous sulfate 160 mg

INTERVENTIONS:
Dietary Supplement: ferrous sulfate 80 mg — 1 tablet per day
  Arms: 80 mg
Dietary Supplement: ferrous sulfate 160 mg — 2 tablets per day
  Arms: 160

SUMMARY:
Serum ferritin is a key indicator of body iron stores and is widely used in monitoring iron status. However, oral iron doses can acutely elevate SF levels, potentially biasing assessments of iron stores during supplementation. This study aims to investigate the extent and duration of the acute iron-induced effect on serum ferritin following the administration of a daily iron dose for two months.

ELIGIBILITY:
Inclusion Criteria:

* Low iron stores (SF levels < 30 µg/L),
* no anemia (Hb > 120 g/L)
* no inflammation (CRP < 5 mg/L)
* 18 to 45 years old.
* Body weight <70 kg
* Normal body Mass Index (18.5-26.5 kg/m2)

Exclusion Criteria:

* Any chronic or acute disease
* Consumption of mineral and vitamin supplements since screening and over the study period
* Blood transfusion, blood donation or significant blood loss over the past 4 months,
* Pregnant or breastfeeding,
* Continuous/long-term use of medication during the whole studies (except for contraceptives)
* Therapeutic iron infusion over the past 6 months,
* Known hypersensitivity or allergy to iron supplements,
* Intention to become pregnant over the course of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum ferritin | Study day 31
  Serum ferritin concentration
Serum ferritin | Study day 37
  Serum ferritin concentration
Serum ferritin | Study day 68
  Serum ferritin concentration
Serum ferritin | Study day 74
  Serum ferritin concentration

SECONDARY OUTCOMES:
alpha(1)-acid-glycoprotein | Study day 1
  alpha(1)-acid-glycoprotein concentration in serum
Serum ferritin | Study day 30
  Serum ferritin concentration
Serum ferritin | Study day 67
  Serum ferritin concentration
Serum ferritin | Study day 20
  Serum ferritin concentration
Serum ferritin | Study day 36
  Serum ferritin concentration
Serum ferritin | Study day 57
  Serum ferritin concentration
Serum ferritin | Study day 72
  Serum ferritin concentration
Serum ferritin | Study day 71
  Serum ferritin concentration
Serum ferritin | Study day 70
  Serum ferritin concentration
Serum ferritin | Study day 69
  Serum ferritin concentration
Serum ferritin | Study day 73
  Serum ferritin concentration
Serum ferritin | Study day 47
  Serum ferritin concentration
Serum ferritin | Study day 35
  Serum ferritin concentration
Serum ferritin | Study day 34
  Serum ferritin concentration
Serum ferritin | Study day 33
  Serum ferritin concentration
Serum ferritin | Study day 32
  Serum ferritin concentration
Serum ferritin | Study day 10
  Serum ferritin concentration
Serum ferritin | Study day 6
  Serum ferritin concentration
Serum ferritin | Study day 3
  Serum ferritin concentration
Serum Ferritin | Study Day 1
  Serum Ferritin concentration
Hemoglobin | Study day 1
  Hemoglobin concentration
C-reactive protein | Study day 1
  C-reactive protein concentration in serum
C-reactive protein | Study day 3
  C-reactive protein concentration in serum
C-reactive protein | Study day 6
  C-reactive protein concentration in serum
C-reactive protein | Study day 10
  C-reactive protein concentration in serum
C-reactive protein | Study day 20
  C-reactive protein concentration in serum
C-reactive protein | Study day 30
  C-reactive protein concentration in serum
C-reactive protein | Study day 31
  C-reactive protein concentration in serum
C-reactive protein | Study day 32
  C-reactive protein concentration in serum
C-reactive protein | Study day 33
  C-reactive protein concentration in serum
C-reactive protein | Study day 34
  C-reactive protein concentration in serum
C-reactive protein | Study day 35
  C-reactive protein concentration in serum
C-reactive protein | Study day 36
  C-reactive protein concentration in serum
C-reactive protein | Study day 37
  C-reactive protein concentration in serum
C-reactive protein | Study day 47
  C-reactive protein concentration in serum
C-reactive protein | Study day 57
  C-reactive protein concentration in serum
C-reactive protein | Study day 67
  C-reactive protein concentration in serum
C-reactive protein | Study day 68
  C-reactive protein concentration in serum
C-reactive protein | Study day 69
  C-reactive protein concentration in serum
C-reactive protein | Study day 70
  C-reactive protein concentration in serum
C-reactive protein | Study day 71
  C-reactive protein concentration in serum
C-reactive protein | Study day 72
  C-reactive protein concentration in serum
C-reactive protein | Study day 73
  C-reactive protein concentration in serum
C-reactive protein | Study day 74
  C-reactive protein concentration in serum
alpha(1)-acid-glycoprotein | Study day 3
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 6
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 10
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 20
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 30
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 31
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 32
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 33
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 34
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 35
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 36
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 37
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 47
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 57
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 67
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 68
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 69
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 70
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 71
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 72
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 73
  alpha(1)-acid-glycoprotein concentration in serum
alpha(1)-acid-glycoprotein | Study day 74
  alpha(1)-acid-glycoprotein concentration in serum
Hemoglobin | Study day 10
  Hemoglobin concentration
Hemoglobin | Study day 20
  Hemoglobin concentration
Hemoglobin | Study day 30
  Hemoglobin concentration
Hemoglobin | Study day 37
  Hemoglobin concentration
Hemoglobin | Study day 47
  Hemoglobin concentration
Hemoglobin | Study day 57
  Hemoglobin concentration
Hemoglobin | Study day 67
  Hemoglobin concentration
Hemoglobin | Study day 74
  Hemoglobin concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Nutrition and Metabolic Epigenetics, Zurich, Canton of Zurich, Switzerland